CLINICAL TRIAL: NCT06841679
Title: A Multi-national, Open-label, Randomized Phase II/III Clinical Study of Utidelone Capsule (UTD2) Combined With Fluoropyrimidine- and Platinum-containing Therapy in First-line Treatment of Patients With Locally Advanced or Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: Utidelone Capsule Combined With Fluoropyrimidine- and Platinum-containing Therapy in First-line Treatment of Patients With Gastric or Gastroesophageal Junction Adenocarcinoma
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Beijing Biostar Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BG02-2404
Record Dates: First submitted 2025-02-10; First posted 2025-02-24 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Gastric or Gastroesophageal Junction Adenocarcinoma
Keywords: UTD2; GC; GEJ
MeSH Terms: interventions — Oxaliplatin; Immune Checkpoint Inhibitors; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental): UTD2 40 mg/m2/d, po, qd, d1-5, q3w combined with CAPOX/FOLFOX with or without a PD-1 inhibitor ( tislelizumab, or pembrolizumab, or nivolumab )
  Interventions: Drug: Utidelone Capsule; Drug: Fluoropyrimidine- and Platinum-containing Therapy; Drug: PD-1 inhibitor
- Cohort 2 (Experimental): UTD2 50 mg/m2/d, po, qd, d1-5, q3w combined with CAPOX/FOLFOX with or without a PD-1 inhibitor ( tislelizumab, or pembrolizumab, or nivolumab )
  Interventions: Drug: Utidelone Capsule; Drug: Fluoropyrimidine- and Platinum-containing Therapy; Drug: PD-1 inhibitor
- Cohort 3 (Experimental): UTD2 60 mg/m2/d, po, qd, d1-5, q3w combined with CAPOX/FOLFOX with or without a PD-1 inhibitor ( tislelizumab, or pembrolizumab, or nivolumab )
  Interventions: Drug: Utidelone Capsule; Drug: Fluoropyrimidine- and Platinum-containing Therapy; Drug: PD-1 inhibitor
- Arm A (Experimental): UTD2 po, on d1-5, q3w (dose decided after the phase II) in combination with CAPOX
  Interventions: Drug: Oxaliplatin; Drug: Utidelone Capsule; Drug: Capecitabine
- Arm B (Active Comparator): CAPOX
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: Utidelone Capsule — UTD2 40 mg/m2/d, po, qd, day 1-5, q3w
  Arms: Cohort 1
Drug: Utidelone Capsule — 50 mg/m2/d, po, qd, day 1-5, q3w
  Arms: Cohort 2
Drug: Utidelone Capsule — 60 mg/m2/d, po, qd, day 1-5, q3w
  Arms: Cohort 3
Drug: Fluoropyrimidine- and Platinum-containing Therapy — CAPOX: Capecitabine 1700 mg/m2/d, po, bid, d1-14，q3w, Oxaliplatin 130 mg/m2, iv, d1, q3w. After completing 6 times (18 weeks) of oxaliplatin treatment, the investigator may decide whether to continue oxaliplatin treatment for up to 8 times (24 weeks) based on the participant's benefits and safety.
  FOLFOX: Oxaliplatin 85 mg/m2, iv, d1, q2w. Folinic Acid 400 mg/m2, iv, d1, q2w, 5-FU 400 mg/m2 IV bolus d1 then 5-FU 2400 mg/m2 IV infusion over 46 to 48 hours, q2w. After completing 9 times (18 weeks) of treatment with oxaliplatin combined with folinic acid and 5-FU, the investigator may decide whether to continue FOLFOX treatment for up to 12 times (24 weeks) based on the participant's benefits and safety.
  Arms: Cohort 1; Cohort 2; Cohort 3
Drug: Oxaliplatin — 130 mg/m2/d, iv, day1, q3w, oxaliplatin will be given up to 6 cycles
  Arms: Arm A; Arm B
Drug: Utidelone Capsule — UTD2 po, on d1-5, q3w (dose decided after the phase II)
  Arms: Arm A
Drug: PD-1 inhibitor — Whether to combine a PD-1 inhibitor will depend on the locally approved indications for the PD-1 inhibitor. If the participant's condition meets the locally approved indications for PD-1 inhibitors, the investigator may determine, in accordance with clinical guidelines, that the participant is eligible to receive treatment with UTD2 combined with fluoropyrimidine- and platinum-containing therapy, with or without a PD-1 inhibitor.
  If a PD-1 inhibitor is administered in combination, tislelizumab (200 mg), or pembrolizumab (200 mg), or nivolumab (360 mg), iv, day1, q3w. Alternatively, the investigator may select the dosage and administration cycle of other locally approved PD-1 inhibitors in accordance with the locally approved package inserts. The PD-1 inhibitor will be given up to 2 years.
  Arms: Cohort 1; Cohort 2; Cohort 3
Drug: Capecitabine — Capecitabine 1700 mg/m2/d po, bid, d1-14，q3w
  Arms: Arm A
Drug: Capecitabine — Capecitabine, 2000 mg/m2/d, po, bid, d1-14, q3w
  Arms: Arm B

SUMMARY:
This is a multi-national, open-label, randomized, seamless phase II/III clinical study of UTD2 combined with fluoropyrimidine- and platinum-containing therapy to evaluate the efficacy and safety in patients with locally advanced or metastatic gastric or gastroesophageal junction adenocarcinoma untreated with systemic treatment in advanced setting.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet the following criteria to be eligible for the study:

  1. Sign the informed consent form (ICF) to participate with accordance with GCP, ICH and local regulations and are willing to adhere to the study protocol.
  2. Male and female aged ≥ 18 years as of the date of baseline visit.
  3. Participant must have unresectable locally advanced or metastatic GC or GEJ and have histologically/pathologic confirmed predominant adenocarcinoma. The documentation of GEJ involvement can include biopsy, endoscopy, or imaging.
  4. Phase II Study: No restriction on PD-L1 expression. Phase III study: Participant must have tumor with PD-L1 Combined Positive Score (CPS) < 1 by immunohistochemical (IHC). IHC results from site are acceptable.
  5. Participant must have at least one measurable lesion per RECIST 1.1 criteria.
  6. Participant must not receive previously systemic treatment in the advanced setting. Previously neoadjuvant/adjuvant therapy for GC or GEJ with no progression after 6 months from completion is allowed. Palliative radiotherapy is allowed.
  7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
  8. Participant with adequate hematological function (CTCAE v5.0 Grade ≤ 1) within 1 week before enrollment (based on routine laboratory values at each site) and who have not received recombinant human granulocyte colony-stimulating factor (rhG-CSF) or blood products/erythropoietin (EPO) within 14 days before enrollment.

     * White blood cell count (WBC) ≥ 3.0 × 109/L;
     * Absolute neutrophil count (ANC) ≥ 1.5 × 109/L;
     * Platelet count (PLT) ≥ 100 × 109/L;
     * Hemoglobin (Hb) ≥ 9.0 g/dL.
  9. Participant with adequate liver and renal function (CTCAE v5.0 Grade ≤ 1) within 1 week before enrollment (based on routine laboratory values at each site).

     * Total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN);
     * Alanine aminotransferase (ALT) ≤ 3 × ULN (≤ 5 × ULN in patients with hepatic metastases);
     * Aspartate aminotransferase (AST) ≤ 3 × ULN (≤ 5 × ULN in patients with hepatic metastases);
     * Creatinine clearance (Ccr) ≥ 50 mL/min.
  10. Female Participants of childbearing potential must agree to use highly effective contraceptive methods during the study and within 6 months after the last dose of the investigational product. Female patients of childbearing potential shall have a negative serum or urine pregnancy test at screening and be willing to have additional pregnancy tests as required throughout the study. Women of non-childbearing potential (WONCBP) must not donate ova from signing informed consent until at least 6 months after the last administration of the investigational product. Please refer to Appendix 1. Males must be surgically sterile (> 6 months since vasectomy with confirmation of no viable sperm), or if engaged in sexual relations (intercourse) with a WOCBP, either his partner must be surgically sterile (eg, hysterectomy, bilateral salpingectomy, bilateral oophorectomy), or an acceptable, highly effective contraceptive method must be used from Screening until 6 months after last IMP administration; or Males with same-sex partners (abstinence from penile-vaginal intercourse) or who are abstinent from heterosexual intercourse are not required to use contraception when this is their preferred and usual lifestyle; or Males must not donate sperm from the first dose of IMP until at least 90 days after the last dose of IMP.

Exclusion Criteria:

* Participants will be excluded from the study for any of the following reasons:

  1. Known HER2-positive tumor (HER2-positive is defined as having an IHC score of 3 +, or IHC2 + and positive HER2 expression by in situ hybridization (ISH) (refer to ASCO/CAP guidelines 2020).
  2. Participants with other malignancies over the past 5 years, except for cured skin basal cell carcinoma, in-situ carcinoma of the cervix, or papillary thyroid cancer.
  3. Participants who have received radiotherapy or other investigational drug or investigational therapy within 4 weeks prior to the first dose of investigational product.
  4. Participants who have undergone major surgery (except biopsy) had significant trauma within 4 weeks prior to the first dose of investigational product or required elective surgery during the study.
  5. Participants with pre-existing > Grade 1 peripheral sensory neuropathy (NCI CTCAE 5.0).
  6. Participants with known hypersensitivity to any components of the investigational product.
  7. Participants who are pregnant (positive pregnancy test) or lactating.
  8. Adverse events due to previous anti-tumor therapy have not recovered to CTCAE v5.0 Grade ≤ 1 (except for alopecia and other toxicities judged by the investigator to have no safety risk).
  9. Participants with esophageal obstruction, pyloric obstruction, intestinal obstruction, or inability to eat on their own after gastrointestinal resection, or other factors that cause difficulty swallowing and inability to take oral drugs.
  10. Participants with symptomatic/uncontrollable central nervous system metastases or meningeal metastases, including but not limited to those with confirmed metastatic disease progression by examination within 2 months after radiotherapy or other local treatment, or who are ineligible for enrollment as judged by the investigator.
  11. Participants with uncontrollable bone metastases, i.e., existing or recent fracture risk, recent need for surgery or local radiotherapy, or other crisis conditions as judged by the investigator.
  12. Participants with uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage (once monthly or more frequently).
  13. Participants with an active infection and who currently require systematic anti-infective therapy.
  14. Participants with known history of human immunodeficiency virus (HIV) infection with an exception that if they have not had an opportunistic infection within the past 12 months, they are eligible.
  15. Participants who are HBV DNA positive or HCV RNA positive (who are HBsAg negative, or HCV antibody negative could be eligible without testing for HBV DNA or HCV RNA).
  16. Participants with a history of severe cardiovascular and cerebrovascular diseases, including but not limited to:

      * Patients with severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmia requiring clinical intervention or second/third-degree atrioventricular block; patients with a mean corrected QT interval (QTcF) > 470 msec obtained from three 12-lead electrocardiograms (ECGs) at rest.
      * Patients who have had an acute coronary syndrome, congestive heart failure, aortic dissection, stroke, or other Grade ≥ 3 cardio-cerebrovascular events within 3 months before the first dose.
      * Patients with clinically uncontrollable hypertension.
      * Symptomatic Cerebral Infarction
      * Patients with other cardiac disorders that put the patients at a high risk as judged by the investigator.
  17. Participants with uncontrolled diabetes mellitus.
  18. Participants with a mental disorder or poor compliance.
  19. Participants also participate in another interventional clinical study or receive other study treatments (patients who have discontinued other investigational treatments and are only in the follow-up period are allowed to be enrolled in this study).
  20. Participants requiring concomitant use of strong CYP3A4 inhibitors or inducers or medications that prolong the QT interval within 14 days prior to the first dose of study treatment and during the study.
  21. Participants with a history of other systemic severe diseases or abnormal laboratory findings that would, in the Investigator's judgment, be inappropriate for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 778 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2030-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of UTD2 and capecitabine in combination with oxaliplatin in Phase II | From Day 1 to Day 21
  dose limiting toxicity (DLT), defined as any toxicity meeting the criteria outlined in the protocol during Cycle 1 in a 21-days cycle
Overall Survival (OS) | 12 months
  From the first dosing until death (from any cause), follow-up began after the end of treatment

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 12 months
  Response rate is the proportion of evaluable patients who are evaluated as having a CR or PR.
Progression Free Survival (PFS) | 12 months
  refers to the time from first dosing to the occurrence of tumor progression or death (whichever occurs first)
Maximum (or peak) serum concentration (Cmax) | 12 months
  Cmax of Utidelone Capsule
Time to peak drug concentration (Tmax) | 12 months
  Tmax of Utidelone Capsule
the area under the concentration-time curve from dosing (time 0) to time t (AUC0-t) | 12 months
  the AUC0-t of Utidelone Capsule
the area under the concentration-time curve from time zero to infinity (AUCinf) | 12 months
  the AUC0inf of Utidelone Capsule
the time required for plasma concentration of a drug to decrease by 50% (t1/2) | 12 months
  the t1/2 of Utidelone Capsule
Treatment-emergent Adverse Events (TEAE) | Until 28 days after the last dose of treatment
  Adverse events (AEs) will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Event version 5.0 (CTCAE v5.0)

OTHER OUTCOMES:
Patient reported outcomes (PRO) | 12 months
  A questionnaire derived from NCI-PRO-CTCAE version 1.0 will be used to assess patient reported safety

CONTACTS AND LOCATIONS:
Locations (10):
- Bioresearch Partner, Hialeah, Florida, United States
- China (9):
  - AnYang Tumor Hospital, Anyang
  - Sun Yat-sen University Cancer Center, Guangzhou
  - Jinan Municipal Central Hospital, Jinan
  - Shandong First Medical University Affiliated Tumor Hospital, Jinan
  - Liaoning Cancer Hospital, Shenyang
  - Shanxi Cancer Hospital, Taiyuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Henan Cancer Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: No